CLINICAL TRIAL: NCT01661075
Title: Quantification of Balance in Acutely Concussed Athletes, Implications for Return to Play Determination
Brief Title: Quantification of Balance in Acutely Concussed Athletes
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Laurie King, Assistant Profressor of Neurology, Oregon Health and Science University
Other Study IDs: 7419_2
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: mTBI; Concussion; Mild Traumatic Brain Injury
Keywords: mTBI; concussion; mild traumatic brain injury; athlete; college; football; soccer
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mTBI: These individuals will have had an mTBI during their respective collegiate athletic season.
- healthy controls: Recruitment of healthy controls who have not suffered an mTBI for balancing testing.

SUMMARY:
The purpose of this pilot project is to determine whether using inertial sensors placed on the waist during routine clinical balance testing (i.e. Balance Error Scoring System) (BESS), will be a more immediate, objective, reliable and sensitive way to measure and quantify balance deficits in individuals with mild Traumatic Brain Injury (mTBI). The investigators are also trying to observe if the sensors can be used to detect balance recovery after a mTBI.

The investigators hypothesis is that collegiate atheltes with mTBI injury will have different recovery periods between their cognitive testing(IMPACT) and their balance measures.

DETAILED DESCRIPTION:
The purpose of this pilot project is to determine whether using inertial sensors (ipod like device) placed on the waist during routine clinical balance testing (i.e. Balance Error Scoring System (BESS), will be a more immediate, objective, reliable and sensitive way to measure and quantify balance deficits in individuals with mild Traumatic Brain Injury (mTBI). The investigators are also trying to observe if the sensors can be used to detect balance recovery after a mTBI.

The participants will be recruited through the local university's athletic department.

The participants will undergo balance tests from the BESS test while wearing a sensor around their waist.The BESS consists of different balance tests; such as balancing on one leg and tandem standing. The participants will also answer questionnaires about their daily lives and cognitive tests. If the participant has had a mTBI they will complete questionnaires about symptoms from their injury and may perform an additional IMPACT test which is a computerized cognitive tests used by coaches, athletic trainers and managing physicians.

Along with the clinical balance tests and questionnaires, the project will use a small sensor placed on the waist to detect sway during quiet stance. An automatic analysis will occur which will provide us with immediate feedback on how stable the participant is during testing.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate athlete

Exclusion Criteria:

* Not a current collegiate athlete,
* recent orthopedic surgery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Collegiate atheltes
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Instrumented Modified Balance Error Scoring System | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A King, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States